CLINICAL TRIAL: NCT07225972
Title: An Open-Label Prospective Randomized Trial of Family Donor-Derived ADV or CMV CTLs Plus Standard of Care (SOC) vs SOC Alone in Children, Adolescents and Young Adults Following Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) With Refractory ADV or CMV Infection/Viremia
Brief Title: Phase 3 Randomized Trial for Refractory ADV or CMV Infection With Family Matched CTLs and Standard of Care (SOC) vs SOC Alone
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: New York Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NYMC 622
Record Dates: First submitted 2025-11-04; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: CMV; AdV Infection; AdV Reactivation; Adenovirus; Cytomegalovirus Infections
MeSH Terms: conditions — Adenoviridae Infections; Cytomegalovirus Infections

STUDY DESIGN:
Intervention Model Description: This study is a prospective, open-label, randomized trial allocating patients to CTLs+SOC and SOC only at a 2:1 ratio. Patients will be enrolled to two cohorts, Cohort 1, ADV and Cohort 2, CMV. For patients with progressive viremia/disease (PD) in the SOC arm, crossover will be allowed to receive CTLs from an eligible family related donor that has screened positive to the specific viral PepTivator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care Medication (Active Comparator): Patients will receive standard of care antiviral therapy for CMV or ADV at the discretion of the physician.
  Interventions: Drug: Standard of Care Antiviral medications
- Standard of Care Medication plus Cytotoxic T-Lymphocytes (CTLs) (Experimental): Patients will be randomized to receiving standard of care antiviral therapy plus family matched donor derived CTLs.
  Interventions: Drug: Standard of Care Antiviral medications; Biological: Viral CTLs

INTERVENTIONS:
Drug: Standard of Care Antiviral medications — Standard of Care medications will be selected by the treating physician for either ADV (Cohort 1) or CMV (cohort 2)
Biological: Viral CTLs — ADV or CMV family matched CTLs will be administered with SOC medications one every 2 weeks as needed up to 5 infusions
  Arms: Standard of Care Medication plus Cytotoxic T-Lymphocytes (CTLs)

SUMMARY:
Patients with refractory ADV or CMV infection post allogeneic stem cell transplant will be randomized to either Family donor-derived viral specific cytotoxic T lymphocytes (CTLs) plus standard of care (SOC) vs SOC alone.

DETAILED DESCRIPTION:
We hypothesize that Family donor-derived viral specific cytotoxic T lymphocytes (CTLs) manufactured by direct selection utilizing the CliniMACS Prodigy® and Cytokine Capture System® plus standard of care (SOC) vs SOC alone in children, adolescents and young adults (CAYA) following allogeneic hematopoietic stem cell transplantation (HSCT) with medically refractory viral infection/viremia and/or intolerant or resistant to anti-viral antibiotic therapy will be associated with a significantly improved probability of Day +100 (time of onset on study) viral progression free survival (VPFS).

ELIGIBILITY:
Patient Eligibility Cohort 1 (ADV) -Patients with ADV infections (Cohort 1) (pneumonitis, hepatitis, cystitis, and/or colitis) post AlloHSCT with one or more of the following: Increasing or persistent ADV RT-PCR DNA (> 1000 ADV PCR copies) after 7 days of appropriate anti-viral therapy AND/OR Medical intolerance to anti-viral therapies including one or more of the following: > grade 2 renal insufficiency secondary to cidofovir and/or other > grade 2 toxicities secondary to cidofovir AND/OR Known resistance to cidofovir

Patient Eligibility (Cohort 2) (CMV)

-Patients with CMV infections (pneumonitis, hepatitis, colitis) with one or more of the following: Increasing or persistent CMV RT-PCR DNA (>1000 copies) after 7 days of appropriate anti-viral therapy AND/OR Medical intolerance to anti-CMV antibiotic therapies: ANC > 500/mm3 secondary to ganciclovir AND/OR > grade 2 renal toxicity secondary to either foscarnet or cidofovir AND/OR Known resistance to ganciclovir and/or foscarnet

* Consent: written informed consent given (by patient or legal representative) prior to any study related procedures
* Performance Status >30% (Lansky < 16 yrs and Karnofsky > 16 years (BOTH COHORTS)
* Age: 0.01 to 30.00 years (BOTH COHORTS)
* Females of childbearing potential with a negative urine pregnancy test at study entry only (BOTH COHORTS)

Donor Eligibility

* Related donor available with a T-cell response to the ADV MACS PepTivators (Cohort 1) or CMV MACS PepTivator (Cohort 2). As defined in Appendix II, B, 8.2, the donor is considered suitable if the percentage of IFN+ T-cells is >0.01% after stimulation with ADV PepTivators (Cohort 1) or CMV PepTivators (Cohort 2).
* Third-party related allogeneic donor: If original donor is not available or does not have a T-cell response to ADV MCAS PepTivator (Cohort 1) or CMV PepTivator (Cohort 2), third party allogeneic donor (family donor > 3 HLA A, B, DR match to recipient) with a T-cell response at least to the ADV MCAS PepTivator (Cohort 1) or CMV PepTivator (Cohort 2) AND
* Allogeneic donor disease screening is complete similar to hematopoietic stem cell donors (Appendix 1) AND
* Obtained informed consents by donor or donor legally authorized representative prior to donor collection

Patient Exclusion Criteria (Both Cohorts)

* Patient with acute GVHD > grade 2 or moderate or extensive chronic GVHD at the time of CTL infusion.
* Patient receiving steroids (>0.5 mg/kg prednisone equivalent) at the time of CTL infusion.
* Patient treated with donor lymphocyte infusion (DLI) within 4 weeks prior to CTL infusion.
* Patient with poor performance status determined by Karnofksy (patients > 16 yrs) or Lansky (patients < 16 years) score < 30%.
* Concomitant enrollment in another experimental clinical trial investigating the treatment of refractory ADV or CMV infections.
* Any known medical condition which cold compromise participation in the study according to investigators assessment.
* Known AIDS or uncontrolled HIV infection
* Known hypersensitivity to iron dextran
* Encephalitis and/or retinitis

Ages: 1 Day to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 69 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2031-12-01 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
Viral PCR to determine resolution of disease | Day 100
  Patients will be monitored weekly by peripheral blood qtPCR values to monitor viral levels for resolution confirmation.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cairo, MD, Principal Investigator — New York Medical College

IPD SHARING:
Plan to Share IPD: No